CLINICAL TRIAL: NCT05539183
Title: Collection of Pleural Effusion Fluid to Design Autologous Onco-immunological Assays
Brief Title: Collection of Pleural Effusion Fluid
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Collaborators: Vrije Universiteit Brussel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 22151PLEUREF
Record Dates: First submitted 2022-08-30; First posted 2022-09-14 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-07

CONDITIONS: Solid Tumor; Pleural Effusion; Metastasis
MeSH Terms: conditions — Pleural Effusion; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Solid cancer patients with malignant pleural effusion (Experimental): Solid cancer patients that have to undergo pleural evacuation because of diagnosed malignant pleural effusion mediated discomfort.
  Interventions: Procedure: Blood withdrawal

INTERVENTIONS:
Procedure: Blood withdrawal — Blood withdrawal

SUMMARY:
At the Laboratory for Molecular and Cellular Therapy (LMCT) of the Vrije Universiteit Brussel, Belgium, we study resistance mechanisms that hamper effective immunotherapy for solid cancer patients. To perform clinically relevant research, we apply autologous human material for functional assessment. The latter requires viable tumor and immune cells.

Solid cancer patients with pleural metastasis often develop pleural effusion. Notably, upon pleural drainage, residual material is obtained that consists of histocompatible tumor and immune cells. Hence with this study, we want to obtain blood and pleural effusion fluid drawn from solid cancer patients with pleural metastases to:

1. Collect, enrich and store primary cells derived from residual pleural effusion fluid and blood at the LMCT (VUB, Belgium)
2. Evaluate characteristics of the cells (phenotype, function,...) and compare content of pleural effusate with blood and clinicopathologic features of the patients.

DETAILED DESCRIPTION:
Malignant pleural effusion (MPE) is characterized by the presence of malignant cells in the pleural cavity and develops in about 15% of patients with malignant disease. Two-thirds of all cases have a pleural effusion as one or sole initial manifestation of malignant disease. Primary tumors that most frequently develop MPE as metastatic disease are lung, breast cancer, and lymphoma accounting for 75% of all cases. Discomforting symptoms of MPE can include chest pain, cough, wheezing, hemoptysis, general discomfort, uneasiness, or ill feeling (malaise), shortness of breath and weight loss. To relief these discomforting symptoms, pleural drainage (evacuation) is routinely performed.

A significant number of solid cancer patients are currently being treated with immunotherapeutic drugs in first or second line or in the framework of a clinical trial. Aside from tumor cell intrinsic mechanisms, we and others previously found that non-malignant tumor infiltrated cells can also install immunotherapy resistance. Hence it remains of utmost importance to study the functional interactions between tumor cells and their non-malignant (solid) micro-environment to increase our current understanding of molecular profiles that predict responsiveness to immunotherapy. By exploiting patient-derived material, we aspire to perform more clinically relevant fundamental and translation research. The primary objective is to collect and compare blood, tumor and MPE-derived cell fractions. The secondary objective is to correlate cellular profiles with clinico-pathologic data.

ELIGIBILITY:
Inclusion Criteria:

* All solid cancer patients with pleural metastases undergoing pleural drainage with available tumor biopsy (upon informed consent)
* >18 years of age

Exclusion Criteria:

* pregnancy

Healthy volunteers will be included for collection of control blood samples (upon informed consent).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Collect and compare blood, tumor and MPE-derived cell fractions | 3 years
  Viable tissue will be processed to single cell suspensions at the research laboratory. Phenotype and function (= description of measurement) will be assessed using flow cytometry and in vitro immune assays (= measurement tools). Specifically we will evaluate the concentration and function of immune cells (derived from blood or pleural effusate like monocytes, macrophages, neutrophils and lymphocytes) and their interaction with autologous tumor cells (only derived from pleural effusate).

SECONDARY OUTCOMES:
Correlate cellular profiles with clinico-pathologic data | 3 years
  We will correlate demographics and biometrical data such as pre-disease history, therapy type, progression free and overall survival and tumor histology with the % of monocytes, macrophages, neutrophils and lymphocytes per patient (obtained from the Primary Outcome Measure). For this purpose, we will use statistical analysis via R software.

CONTACTS AND LOCATIONS:
Overall Officials: Lore Decoster, MD PhD, Principal Investigator — Universitair Ziekenhuis Brussel

IPD SHARING:
Plan to Share IPD: No
Samples will be pseudonymized and processed via RedCAP